CLINICAL TRIAL: NCT01882569
Title: Detection of Immune Changes as a Result of Surgical Trauma in Human Back Surgery Subjects: Optimization of CyTOF Analysis
Brief Title: Optimization of Time-of-Flight Mass Cytometry (CyTOF) Analysis for Evaluation of Immune Changes Following Surgery
Status: Completed | Type: Observational
Sponsor: Martin Angst (Other)
Responsible Party: Sponsor-Investigator, Martin Angst, Professor of Anesthesia, Stanford University
Organization: Stanford University (Other)
Other Study IDs: 24014
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Surgical Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Back surgery

SUMMARY:
Surgical trauma triggers a massive inflammatory response. Over time, both the innate and adaptive branches of the immune system are affected by surgical trauma. The purpose of this study is to use a single cell flow cytometry approach to characterize the cellular and molecular mechanisms involved in the inflammatory response to surgical trauma.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 - 90
2. Men and women
3. Undergo back surgery

Exclusion Criteria:

1. Any systemic disease that might compromise the immune system (e.g. lupus)
2. Current diagnosis of cancer
3. Any condition that, in the opinion of the investigator, might compromise the integrity of the study or safety of the participant.
4. Unwilling to sign informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Generally healthy patients undergoing back surgery
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2012-05; Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Numerical (cell frequencies) and functional (phosphorylation of signaling proteins and transcription factors) changes of all circulating immune cells | Immediately before to surgery, 1 hour after surgery, 24 hours after surgery, and day of hospital discharge
  This is an exploratory study.

CONTACTS AND LOCATIONS:
Overall Officials: Martin S Angst, MD, Principal Investigator — Stanford University SOM
Locations (1):
- Stanford University Hospital, Stanford, California, United States